CLINICAL TRIAL: NCT00344318
Title: To Assess the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Pneumococcal Conjugate Vaccine Compared to Prevenar™, Co-administered With DTPw-HBV/Hib & OPV or IPV Vaccines as a 3-dose Primary Immunization Course During the First 6 Months of Age
Brief Title: Safety and Immunogenicity Study of GlaxoSmithKline (GSK) Biologicals' 10-valent Pneumococcal Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 107007
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-05

CONDITIONS: Infections, Streptococcal
Keywords: Immunogenicity; Safety; Pneumococcal vaccine; Pneumococcal disease
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Tritanrix-HepB vaccine; Hiberix

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (4):
- Synflorix 1 Group (Experimental): Subjects aged 6-12 weeks from the Philippines receiving Synflorix™ vaccine, co-administered with Tritanrix™-HepB/Hiberix™ and Polio Sabin™ vaccines at 6, 10, 14 weeks of age.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: Tritanrix-HepB; Biological: Hiberix; Biological: Polio Sabin.; Biological: Poliorix.
- Synflorix 2 Group (Experimental): Subjects aged 6-12 weeks from Poland receiving Synflorix™ vaccine co-administered with Tritanrix™-HepB/Hiberix™ and Poliorix™ vaccines at 2, 4, 6 months of age.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: Tritanrix-HepB; Biological: Hiberix; Biological: Polio Sabin.; Biological: Poliorix.
- Prevenar 1 Group (Active Comparator): Subjects aged 6-12 weeks from the Philippines receiving the Prevenar™ vaccine, co-administered with Tritanrix™-HepB/Hiberix™ and Polio Sabin™ at 6, 10, 14 weeks of age.
  Interventions: Biological: Prevenar; Biological: Tritanrix-HepB; Biological: Hiberix; Biological: Polio Sabin.; Biological: Poliorix.
- Prevenar 2 Group (Active Comparator): Subjects aged 6-12 weeks from Poland receiving the Prevenar™ vaccine, co-administered with Tritanrix™-HepB/Hiberix™ and Poliorix™ at 2, 4, 6 months of age.
  Interventions: Biological: Prevenar; Biological: Tritanrix-HepB; Biological: Hiberix; Biological: Polio Sabin.; Biological: Poliorix.

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine GSK1024850A — 3 Intramuscular injections.
  Arms: Synflorix 1 Group; Synflorix 2 Group
Biological: Prevenar — 3 Intramuscular injections
  Arms: Prevenar 1 Group; Prevenar 2 Group
Biological: Tritanrix-HepB — 3 Intramuscular injections
  Other Names: DTPw-HBV
Biological: Hiberix — Reconstituted with Tritanrix before injection
  Other Names: Hib
Biological: Polio Sabin. — 3 oral doses.
  Other Names: OPV
Biological: Poliorix. — 3 intramuscular injections
  Other Names: IPV

SUMMARY:
This study will evaluate safety, reactogenicity and immunogenicity of GSK Biologicals' pneumococcal conjugate vaccine compared to Prevenar™ when co-administered with DTPw-HBV/Hib and OPV or IPV vaccines, according to 2 different schedules: 6-10-14 weeks or 2-4-6 months of age.

The study has 2 groups.

* One group of subjects will receive a 3-dose primary vaccination with the GSK Biologicals' pneumococcal conjugate vaccine (three different lots will be used and randomly allocated).
* The 2nd group of subjects will receive a 3-dose primary vaccination with Prevenar™.

All children will receive concomitantly DTPw-HBV/Hib and OPV or IPV vaccines. This protocol posting deals with objectives & outcome measures of the primary study. The objectives & outcome measures of the Booster study are presented in a separate protocol posting (NCT number =00547248).

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007

ELIGIBILITY:
Inclusion Criteria:

* Male or female between, and including, 6-12 weeks (42 to 90 days) of age at the time of the first vaccination.
* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born after a gestation period between 36 and 42 weeks.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting one month before each dose of vaccine(s) and ending 7 days after dose 1 and dose 2 or 1 month after dose 3.
* Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b, and/or S. pneumoniae with the exception of vaccines where the first dose can be given within the first two weeks of life according to the national recommendations
* History of or intercurrent diphtheria, tetanus, pertussis, hepatitis B, polio, and Haemophilus influenzae type b diseases.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of seizures (this criterion does not apply to subjects who have had a single, uncomplicated febrile convulsion in the past) or neurological disease.
* Acute disease at the time of enrolment
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the active phase of the study.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 806 (Actual)
Dates: Start 2006-08-07 (Actual); Primary Completion 2007-04-27 (Actual); Study Completion 2007-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- GSK Investigational Site, City of Muntinlupa, Philippines
- Poland (5):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Tuchola
  - GSK Investigational Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Knuf M, Szenborn L, Moro M, Petit C, Bermal N, Bernard L, Dieussaert I, Schuerman L. Immunogenicity of routinely used childhood vaccines when coadministered with the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S97-S108. doi: 10.1097/INF.0b013e318199f61b. PMID 19325452
- [Derived] Bermal N, Szenborn L, Chrobot A, Alberto E, Lommel P, Gatchalian S, Dieussaert I, Schuerman L. The 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) coadministered with DTPw-HBV/Hib and poliovirus vaccines: assessment of immunogenicity. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S89-96. doi: 10.1097/INF.0b013e318199f901. PMID 19325451
- [Derived] Chevallier B, Vesikari T, Brzostek J, Knuf M, Bermal N, Aristegui J, Borys D, Cleerbout J, Lommel P, Schuerman L. Safety and reactogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) when coadministered with routine childhood vaccines. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S109-18. doi: 10.1097/INF.0b013e318199f62d. PMID 19325447
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 107007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Started | 300 | 303 | 100 | 103
Completed | 296 | 298 | 99 | 100
Not Completed | 4 | 5 | 1 | 3
Not completed — Adverse Event | 0 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 2
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group | Total
Number analyzed (Participants) | 300 | 303 | 100 | 103 | 806
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 7.5 (1.64) | 7.4 (1.5) | 7.4 (1.53) | 7.5 (1.55) | 7.45 (1.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 141 | 48 | 46 | 381
  Male | 154 | 162 | 52 | 57 | 425

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Rectal Temperature Above (>) 39.0 Degrees Celsius (°C)
Description: Fever was measured as rectal temperature. Assessment of occurrences of fever > 39.0 °C was performed post doses 1, 2 and 3 and across doses of Synflorix™ or Prevenar™ vaccine.
Time Frame: Within 4 day (Days 0-3) after each dose and across doses
Population: The analysis was performed on the Total vaccinated cohort, which included all subjects with at least one vaccine administration documented and who had their symptom sheets filled in. For reasons of safety analysis related to rectal temperature, subjects were pooled to form the Synflorix Pooled Group and Prevenar Group.
Measure: Count of Participants; unit: Participants
Groups:
- Synflorix Pooled Group: Synflorix 1 Group and Synflorix 2 Group pooled together
- Prevenar Pooled Group: Prevenar 1 Group and Prevenar 2 Group pooled together
Arm/Group | Synflorix Pooled Group | Prevenar Pooled Group
Number analyzed (Participants) | 599 | 199
Participants
  Fever > 39.0°C, post Dose 1: number analyzed (Participants) | 598 | 199
  Fever > 39.0°C, post Dose 1 | 31 | 6
  Fever > 39.0°C, post Dose 2: number analyzed (Participants) | 594 | 199
  Fever > 39.0°C, post Dose 2 | 30 | 13
  Fever > 39.0°C, post Dose 3 | 42 | 8
  Fever > 39.0°C, across doses | 88 | 23
Statistical Analysis 1: Comparison: Synflorix Pooled Group vs Prevenar Pooled Group; Analysis aimed to demonstrate that Synflorix™ vaccine administered as a 3-dose primary vaccination course (either at 6-10-14 weeks or at 2-4-6 months of age), is non-inferior to Prevenar™ in terms of the incidence of post-immunization rectal fever >39.0°C, when co-administered with Tritanrix™-HepB/Hiberix™ and Polio Sabin™ or Poliorix™ vaccines; Test type: Non-Inferiority or Equivalence — Standardized asymptotic 95% confidence interval (CI) for the difference [Synflorix™ minus Prevenar™] in terms of percentages of subjects reporting rectal fever >39.0°C after Dose 1 was computed; Difference in percentage = 2.17, 95% CI 2-sided [-1.51 to 4.88]
Statistical Analysis 2: Comparison: Synflorix Pooled Group vs Prevenar Pooled Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Towards this, standardized asymptotic 95% confidence interval (CI) for the difference [Synflorix™ minus Prevenar™] in terms of percentages of subjects reporting rectal fever >39.0°C after Dose 2 was computed; Difference in percentage = -1.48, 95% CI [-6.05 to 1.92]
Statistical Analysis 3: Comparison: Synflorix Pooled Group vs Prevenar Pooled Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Towards this, standardized asymptotic 95% confidence interval (CI) for the difference [Synflorix™ minus Prevenar™] in terms of percentages of subjects reporting rectal fever >39.0°C after Dose 3 was computed; Difference in percentage = 3.05, 95% CI 2-sided [-1.02 to 6.19]
Statistical Analysis 4: Comparison: Synflorix Pooled Group vs Prevenar Pooled Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Standardized asymptotic 95% confidence interval (CI) for the difference [Synflorix™ minus Prevenar™] in terms of percentages of subjects reporting rectal fever >39.0°C across doses was computed; Difference in percentage = 3.13, 95% CI 2-sided [-2.65 to 8.01]

2. Secondary Outcome: Number of Subjects With Any and Any Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Grade 3 pain was defined as crying when limb was moved/spontaneously painful. Grade 3 swelling/redness was defined as swelling/redness larger than (>) 30 millimeters (mm). "Any" is defined as incidence of the specified symptom regardless of intensity.
Time Frame: Within 4 day (Days 0-3) after each dose and across doses
Population: The analysis was performed on the Total vaccinated cohort, which included all subjects with at least one vaccine administration documented and who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 299 | 300 | 99 | 100
Participants
  Any Pain, Post Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  Any Pain, Post Dose 1 | 240 | 206 | 76 | 65
  Grade 3 Pain, Post Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  Grade 3 Pain, Post Dose 1 | 52 | 59 | 19 | 17
  Any Redness, Post Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  Any Redness, Post Dose 1 | 126 | 199 | 35 | 65
  Grade 3 Redness, Post Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  Grade 3 Redness, Post Dose 1 | 10 | 30 | 6 | 8
  Any Swelling, Post Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  Any Swelling, Post Dose 1 | 142 | 153 | 39 | 56
  Grade 3 Swelling, Post Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  Grade 3 Swelling, Post Dose 1 | 41 | 43 | 15 | 9
  Any Pain, Post Dose 2: number analyzed (Participants) | 296 | 299 | 99 | 100
  Any Pain, Post Dose 2 | 191 | 186 | 55 | 61
  Grade 3 Pain, Post Dose 2: number analyzed (Participants) | 296 | 299 | 99 | 100
  Grade 3 Pain, Post Dose 2 | 18 | 31 | 8 | 12
  Any Redness, Post Dose 2: number analyzed (Participants) | 296 | 299 | 99 | 100
  Any Redness, Post Dose 2 | 135 | 204 | 44 | 59
  Grade 3 Redness, Post Dose 2: number analyzed (Participants) | 296 | 299 | 99 | 100
  Grade 3 Redness, Post Dose 2 | 8 | 9 | 1 | 2
  Any Swelling, Post Dose 2: number analyzed (Participants) | 296 | 299 | 99 | 100
  Any Swelling, Post Dose 2 | 98 | 163 | 29 | 51
  Grade 3 Swelling, Post Dose 2: number analyzed (Participants) | 296 | 299 | 99 | 100
  Grade 3 Swelling, Post Dose 2 | 27 | 19 | 5 | 5
  Any Pain, Post Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  Any Pain, Post Dose 3 | 168 | 173 | 44 | 56
  Grade 3 Pain, Post Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  Grade 3 Pain, Post Dose 3 | 14 | 23 | 1 | 8
  Any Redness, Post Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  Any Redness, Post Dose 3 | 158 | 209 | 45 | 70
  Grade 3 Redness, Post Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  Grade 3 Redness, Post Dose 3 | 3 | 8 | 0 | 4
  Any Swelling, Post Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  Any Swelling, Post Dose 3 | 84 | 151 | 25 | 53
  Grade 3 Swelling, Post Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  Grade 3 Swelling, Post Dose 3 | 15 | 19 | 4 | 10
  Any Pain, Across Doses | 258 | 255 | 82 | 89
  Grade 3 Pain, Across Doses | 64 | 83 | 22 | 25
  Any Redness, Across Doses | 221 | 265 | 67 | 90
  Grade 3 Redness, Across Doses | 18 | 42 | 6 | 12
  Any Swelling, Across Doses | 174 | 226 | 42 | 75
  Grade 3 Swelling, Across Doses | 57 | 65 | 16 | 16

3. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever (defined as rectal temperature ≥ 38.0°C), irritability, and loss of appetite. Grade 3 (G3) drowsiness was defined as drowsiness which prevented normal everyday activities. Grade 3 (G3) fever was defined as fever (rectal temperature) above (>) 40.0 degree Celsius (°C). Grade 3 (G3) irritability was defined as crying that could not be comforted/preventing normal activity. Grade 3 (G3) loss of appetite was defined as the subject not eating at all. "Any" is defined as incidence of the specified symptom regardless of intensity or relationship to study vaccination. Related (REL) = Symptom assessed by the investigator as causally related to vaccination.
Time Frame: Within 4-day (Days 0-3) after each dose and across doses
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 299 | 300 | 99 | 100
Participants
  Any Drowsiness, Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  Any Drowsiness, Dose 1 | 154 | 223 | 45 | 75
  G3 Drowsiness, Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  G3 Drowsiness, Dose 1 | 6 | 10 | 3 | 1
  REL Drowsiness Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  REL Drowsiness Dose 1 | 154 | 222 | 45 | 75
  Any Fever, Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  Any Fever, Dose 1 | 214 | 190 | 74 | 54
  G3 Fever, Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  G3 Fever, Dose 1 | 0 | 0 | 0 | 0
  REL Fever, Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  REL Fever, Dose 1 | 214 | 190 | 74 | 54
  Any Irritability, Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  Any Irritability, Dose 1 | 236 | 269 | 78 | 83
  G3 Irritability, Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  G3 Irritability, Dose 1 | 11 | 60 | 3 | 17
  REL Irritability, Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  REL Irritability, Dose 1 | 236 | 266 | 78 | 83
  Any Loss of appetite, Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  Any Loss of appetite, Dose 1 | 104 | 166 | 26 | 52
  G3 Loss of appetite, Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  G3 Loss of appetite, Dose 1 | 1 | 1 | 1 | 1
  REL Loss of appetite, Dose 1: number analyzed (Participants) | 299 | 299 | 99 | 100
  REL Loss of appetite, Dose 1 | 104 | 165 | 26 | 51
  Any Drowsiness, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  Any Drowsiness, Dose 2 | 102 | 172 | 25 | 57
  G3 Drowsiness, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  G3 Drowsiness, Dose 2 | 1 | 9 | 1 | 2
  REL Drowsiness, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  REL Drowsiness, Dose 2 | 102 | 172 | 24 | 56
  Any Fever, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  Any Fever, Dose 2 | 182 | 184 | 63 | 51
  G3 Fever, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  G3 Fever, Dose 2 | 0 | 0 | 0 | 0
  REL Fever, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  REL Fever, Dose 2 | 182 | 184 | 63 | 50
  Any Irritability, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  Any Irritability, Dose 2 | 185 | 238 | 49 | 73
  G3 Irritability, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  G3 Irritability, Dose 2 | 8 | 37 | 3 | 9
  REL Irritability, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  REL Irritability, Dose 2 | 185 | 237 | 48 | 72
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  Any Loss of appetite, Dose 2 | 66 | 117 | 20 | 28
  G3 Loss of appetite, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  G3 Loss of appetite, Dose 2 | 0 | 0 | 0 | 0
  REL Loss of appetite, Dose 2: number analyzed (Participants) | 296 | 298 | 99 | 100
  REL Loss of appetite, Dose 2 | 66 | 116 | 19 | 27
  Any Drowsiness, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  Any Drowsiness, Dose 3 | 90 | 152 | 25 | 41
  G3 Drowsiness, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  G3 Drowsiness, Dose 3 | 2 | 5 | 0 | 0
  REL Drowsiness, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  REL Drowsiness, Dose 3 | 90 | 151 | 25 | 40
  Any Fever, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  Any Fever, Dose 3 | 147 | 163 | 50 | 49
  G3 Fever, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  G3 Fever, Dose 3 | 0 | 0 | 0 | 1
  REL Fever, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  REL Fever, Dose 3 | 147 | 162 | 50 | 49
  Any Irritability, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  Any Irritability, Dose 3 | 169 | 225 | 43 | 64
  G3 Irritability, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  G3 Irritability, Dose 3 | 7 | 22 | 1 | 2
  REL Irritability, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  REL Irritability, Dose 3 | 169 | 223 | 43 | 64
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  Any Loss of appetite, Dose 3 | 61 | 113 | 19 | 19
  G3 Loss of appetite, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  G3 Loss of appetite, Dose 3 | 1 | 1 | 0 | 0
  REL Loss of appetite, Dose 3: number analyzed (Participants) | 296 | 298 | 99 | 100
  REL Loss of appetite, Dose 3 | 61 | 113 | 19 | 19
  Any Drowsiness, Across Doses | 184 | 256 | 56 | 85
  G3 Drowsiness, Across Doses | 9 | 17 | 3 | 3
  REL Drowsiness, Across Doses | 184 | 256 | 56 | 85
  Any Fever, Across Doses | 255 | 261 | 88 | 77
  G3 Fever, Across Doses | 0 | 0 | 0 | 1
  REL Fever, Across Doses | 255 | 261 | 88 | 77
  Any Irritability, Across Doses | 258 | 289 | 82 | 93
  G3 Irritability, Across Doses | 22 | 89 | 6 | 24
  REL Irritability, Across Doses | 258 | 289 | 82 | 93
  Any Loss of appetite, Across | 140 | 221 | 39 | 64
  G3 Loss of appetite, Across | 1 | 2 | 1 | 1
  REL Loss of appetite, Across | 140 | 220 | 39 | 63

4. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" is defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: Within 31 days (Days 0-30) after each vaccination
Population: The analysis was performed on the Total vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 300 | 303 | 100 | 103
Participants | 168 | 166 | 46 | 61

5. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the Active Phase: From Month 0 to Month 3 for Synflorix 1 Group and Prevenar 1 Group and from Month 0 to Month 5 for the Synflorix 2 Group and Prevenar 2 Group
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 300 | 303 | 100 | 103
Participants | 6 | 34 | 1 | 9

6. Secondary Outcome: Number of Subjects With Serious Adverse (SAEs)
Description: as for outcome 5
Time Frame: During the Extended Safety Follow-Up Phase: At Month 8 for Synflorix 1 Group and Prevenar 1 Group and at Month 10 for the Synflorix 2 Group and Prevenar 2 Group
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 300 | 303 | 100 | 103
Participants | 16 | 52 | 4 | 19

7. Secondary Outcome: Concentrations of Antibodies Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F
Description: Seropositivity status, defined as Anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations ≥ 0.05 microgram per milliliter (µg/mL).
Time Frame: One month after the administration of the 3rd vaccine dose of Synflorix™ and Prevenar™
Population: The analysis was performed on the According-To-Protocol (ATP) Cohort for immunogenecity, which included all evaluable subjects whith available immunogenecity data. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 285 | 285 | 95 | 96
μg/mL
  Anti-1 POST: number analyzed (Participants) | 285 | 285 | 94 | 96
  Anti-1 POST | 3.23 [2.94 to 3.54] | 1.04 [0.94 to 1.15] | 0.03 [0.03 to 0.4] | 0.03 [0.03 to 0.03]
  Anti-4 POST | 4.96 [4.46 to 5.51] | 1.64 [1.49 to 1.8] | 5.68 [4.94 to 6.53] | 2.14 [1.88 to 2.44]
  Anti-5 POST | 4.87 [4.5 to 5.26] | 1.62 [1.48 to 1.78] | 0.03 [0.03 to 0.04] | 0.03 [0.03 to 0.03]
  Anti-6B POST | 1.19 [1.02 to 1.38] | 0.73 [0.64 to 0.84] | 1.06 [0.8 to 1.4] | 1.23 [0.96 to 1.58]
  Anti-7F POST | 4.84 [4.45 to 5.27] | 2.25 [2.07 to 2.45] | 0.05 [0.04 to 0.06] | 0.04 [0.03 to 0.04]
  Anti-9V POST | 4.04 [3.66 to 4.46] | 1.51 [1.37 to 1.66] | 5.07 [4.32 to 5.96] | 2.7 [2.32 to 3.14]
  Anti-14 POST | 6.45 [5.65 to 7.38] | 3.31 [2.98 to 3.68] | 5.88 [4.71 to 7.34] | 5.23 [4.39 to 6.24]
  Anti-18C POST | 11.56 [10.22 to 13.08] | 3.74 [3.28 to 4.28] | 3.71 [3.14 to 4.38] | 2.64 [2.25 to 3.11]
  Anti-19F POST | 10.46 [9.32 to 11.74] | 5.3 [4.77 to 5.89] | 4.68 [4.02 to 5.45] | 2.38 [2.04 to 2.78]
  Anti-23F POST | 2.23 [1.98 to 2.5] | 1.11 [0.98 to 1.26] | 2.28 [1.7 to 3.06] | 2.2 [1.83 to 2.65]

8. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations Equal to or Above (≥) 0.2 Microgram Per Milliliter (µg/mL)
Description: Cut-off values assessed were greater than or equal to 0.2 microgram per milliliter (µg/mL) in the sera of subjects.
Time Frame: One month after the administration of the 3rd vaccine dose of Synflorix™ and Prevenar™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 285 | 285 | 95 | 96
Participants
  Anti-1 POST: number analyzed (Participants) | 285 | 285 | 94 | 96
  Anti-1 POST | 285 | 280 | 3 | 3
  Anti-4 POST | 283 | 282 | 95 | 96
  Anti-5 POST | 285 | 282 | 3 | 2
  Anti-6B POST | 260 | 244 | 82 | 91
  Anti-7F POST | 284 | 285 | 9 | 5
  Anti-9V POST | 284 | 285 | 95 | 96
  Anti-14 POST | 285 | 285 | 95 | 96
  Anti-18C POST | 284 | 281 | 95 | 95
  Anti-19F POST | 285 | 282 | 94 | 95
  Anti-23F POST | 277 | 269 | 90 | 95

9. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations Equal to or Above (≥) 0.05 Microgram Per Liter (µg/mL)
Description: Cut-off values assessed were greater than or equal to 0.05 microgram per liter (µg/mL) in the sera of subjects.
Time Frame: One month after the administration of the 3rd vaccine dose of Synflorix™ and Prevenar™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 285 | 285 | 95 | 96
Participants
  Anti-1 POST: number analyzed (Participants) | 285 | 285 | 94 | 96
  Anti-1 POST | 285 | 285 | 20 | 13
  Anti-4 POST | 285 | 285 | 95 | 96
  Anti-5 POST | 285 | 285 | 19 | 13
  Anti-6B POST | 279 | 274 | 92 | 91
  Anti-7F POST | 285 | 285 | 37 | 22
  Anti-9V POST | 285 | 285 | 95 | 96
  Anti-14 POST | 285 | 285 | 95 | 96
  Anti-18C POST | 284 | 285 | 95 | 95
  Anti-19F POST | 285 | 285 | 95 | 95
  Anti-23F POST | 285 | 279 | 91 | 96

10. Secondary Outcome: Opsonophagocytic Activity (OPA) Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F
Description: Seropositivity status, defined as Opsonophagocytic activity against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F ≥ 8
Time Frame: One month after the administration of the 3rd vaccine dose of Synflorix™ and Prevenar™
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 142 | 145 | 46 | 49
Titers
  OPA Anti-1: number analyzed (Participants) | 142 | 144 | 46 | 49
  OPA Anti-1 | 93.7 [68.2 to 128.7] | 14.8 [11.2 to 19.6] | 4.2 [3.8 to 4.5] | 4 [4 to 4]
  OPA Anti-4: number analyzed (Participants) | 138 | 145 | 43 | 49
  OPA Anti-4 | 1008.7 [849.1 to 1198.4] | 602.9 [494.8 to 734.6] | 1229.9 [975.5 to 1550.7] | 513 [388.2 to 677.9]
  OPA Anti-5: number analyzed (Participants) | 140 | 144 | 46 | 49
  OPA Anti-5 | 209.3 [176.6 to 248] | 67.2 [52.2 to 86.6] | 4 [4 to 4] | 4 [4 to 4]
  OPA Anti-6B: number analyzed (Participants) | 142 | 145 | 43 | 49
  OPA Anti-6B | 963.5 [714.7 to 1299] | 361.9 [255 to 513.7] | 1762.2 [975.3 to 3184] | 805 [436.9 to 1483.4]
  OPA Anti-7F: number analyzed (Participants) | 137 | 144 | 44 | 49
  OPA Anti-7F | 5196.4 [4349.2 to 6208.6] | 2002.2 [1543.1 to 2597.9] | 14.2 [6.9 to 29.4] | 6.9 [4.3 to 11.1]
  OPA Anti-9V: number analyzed (Participants) | 130 | 144 | 43 | 49
  OPA Anti-9V | 1631.9 [1343.8 to 1981.9] | 1171.7 [966.1 to 1421.1] | 1713.3 [1294.6 to 2267.5] | 1166 [782.6 to 1737.2]
  OPA Anti-14 | 1669.1 [1267.7 to 2197.6] | 640 [520.2 to 787.5] | 2117.4 [1210.9 to 3702.6] | 947.6 [658.6 to 1363.4]
  OPA Anti-18C: number analyzed (Participants) | 139 | 144 | 45 | 49
  OPA Anti-18C | 673.3 [569.7 to 795.8] | 174.9 [137.1 to 223.1] | 283.7 [209.6 to 384.1] | 127 [86.4 to 186.5]
  OPA Anti-19F: number analyzed (Participants) | 139 | 143 | 46 | 49
  OPA Anti-19F | 1121.7 [931.5 to 1350.6] | 337.8 [262.9 to 434.1] | 81.6 [53 to 125.5] | 35.9 [25.7 to 50.1]
  OPA Anti-23F: number analyzed (Participants) | 141 | 143 | 43 | 49
  OPA Anti-23F | 2186.6 [1845.4 to 2590.9] | 920.6 [678 to 1249.9] | 4126.6 [2609 to 6526.8] | 3895.4 [2842.8 to 5337.8]

11. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity (OPA) Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Equal to or Above (≥) 8
Description: Seropositivity status, defined as Opsonophagocytic activity against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C , 19F and 23F ≥ 8.
Time Frame: One month after the administration of the 3rd vaccine dose of Synflorix™ and Prevenar™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 142 | 145 | 46 | 49
Participants
  OPA Anti-1: number analyzed (Participants) | 142 | 144 | 46 | 49
  OPA Anti-1 | 117 | 62 | 1 | 0
  OPA Anti-4: number analyzed (Participants) | 138 | 145 | 43 | 49
  OPA Anti-4 | 137 | 143 | 43 | 49
  OPA Anti-5: number analyzed (Participants) | 140 | 144 | 46 | 49
  OPA Anti-5 | 139 | 127 | 0 | 0
  OPA Anti-6B: number analyzed (Participants) | 142 | 145 | 43 | 49
  OPA Anti-6B | 132 | 122 | 40 | 44
  OPA Anti-7F: number analyzed (Participants) | 137 | 144 | 44 | 49
  OPA Anti-7F | 137 | 141 | 10 | 5
  OPA Anti-9V: number analyzed (Participants) | 130 | 144 | 43 | 49
  OPA Anti-9V | 130 | 144 | 43 | 49
  OPA Anti-14 | 138 | 142 | 43 | 48
  OPA Anti-18C: number analyzed (Participants) | 139 | 144 | 45 | 49
  OPA Anti-18C | 138 | 137 | 45 | 48
  OPA Anti-19F: number analyzed (Participants) | 139 | 143 | 46 | 49
  OPA Anti-19F | 137 | 142 | 42 | 45
  OPA Anti-23F: number analyzed (Participants) | 141 | 143 | 43 | 49
  OPA Anti-23F | 141 | 132 | 42 | 49

12. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: Seropositivity status, defined as Anti-pneumococcal cross-reactive serotypes 6A and 19A antibody concentrations ≥ 0.05 microgram per milliliter (µg/mL).
Time Frame: One month after the administration of the 3rd vaccine dose of Synflorix™ and Prevenar™
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 285 | 285 | 95 | 96
μg/mL
  Anti-6A | 0.3 [0.26 to 0.35] | 0.17 [0.15 to 0.2] | 0.23 [0.18 to 0.3] | 0.26 [0.2 to 0.33]
  Anti-19A: number analyzed (Participants) | 285 | 284 | 95 | 96
  Anti-19A | 0.36 [0.31 to 0.41] | 0.29 [0.25 to 0.34] | 0.18 [0.15 to 0.22] | 0.12 [0.1 to 0.15]

13. Secondary Outcome: Number of Subjects With Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A Equal to or Above (≥) 0.05 Microgram Per Milliliter (μg/mL)
Description: Cut-off values assessed were greater than or equal to 0.05 microgram per milliliter (μg/mL) in the sera of subjects seronegative before vaccination.
Time Frame: One month after the administration of the 3rd vaccine dose of Synflorix™ and Prevenar™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 285 | 285 | 95 | 96
Participants
  Anti-6A | 261 | 230 | 84 | 84
  Anti-19A: number analyzed (Participants) | 285 | 284 | 95 | 96
  Anti-19A | 169 | 164 | 90 | 83

14. Secondary Outcome: Opsonophagocytic Activity (OPA) Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: Seropositivity status, defined as Opsonophagocytic activity against pneumococcal cross-reactive serotypes 6A and 19A ≥ 8
Time Frame: One month after the administration of the 3rd vaccine dose of Synflorix™ and Prevenar™
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 137 | 143 | 44 | 49
Titers
  OPA Anti-6A: number analyzed (Participants) | 127 | 137 | 43 | 48
  OPA Anti-6A | 93.1 [64.1 to 135.2] | 60.5 [40.7 to 89.9] | 137.3 [69.7 to 270.3] | 175.1 [87.2 to 351.6]
  OPA Anti-19A | 10.6 [7.9 to 14.2] | 10.1 [7.8 to 13.1] | 4.2 [3.8 to 4.7] | 4 [4 to 4]

15. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity (OPA) Against Cross-reactive Pneumococcal Serotypes 6A and 19A Equal to or Above (≥) 8
Description: as for outcome 14
Time Frame: One month after the administration of the 3rd vaccine dose of Synflorix™ and Prevenar™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 137 | 143 | 44 | 49
Participants
  OPA Anti-6A: number analyzed (Participants) | 127 | 137 | 43 | 48
  OPA Anti-6A | 91 | 83 | 34 | 36
  OPA Anti-19A | 35 | 41 | 1 | 0

16. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD)
Description: Seropositivity status, defined as Anti-PD antibody concentrations ≥ 100 ELISA units per milliliter ( EL.U/mL)
Time Frame: One month after the administration of the 3rd vaccine dose of Synflorix™ and Prevenar™
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 284 | 285 | 95 | 96
EL.U/mL | 3800 [3481.2 to 4148] | 2002 [1780 to 2251.6] | 105.2 [85.3 to 129.6] | 66.6 [58.5 to 75.8]

17. Secondary Outcome: Number of Subjects With Concentrations of Antibodies Against Protein D (Anti-PD) Equal to or Above (≥) 100 ELISA Units Per Milliliter (EL.U/mL)
Description: Cut-off values assessed were greater than or equal to 100 ELISA units per milliliter (EL.U/mL) in the sera of subjects.
Time Frame: One month after the administration of the 3rd vaccine dose of Synflorix™ and Prevenar™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 284 | 285 | 95 | 96
Participants | 284 | 285 | 39 | 18

18. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration Equal to or Above 0.15 Microgram Per Milliliter (µg/ mL)
Description: Cut-off values assessed were greater than or equal to 0.15 microgram per milliliter (µg/ mL) in the sera of subjects.
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 140 | 140 | 49 | 47
Participants | 140 | 140 | 49 | 47

19. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration Equal to or Above 1.0 Microgram Per Milliliter (µg/mL)
Description: Cut-off values assessed were greater than or equal to 1.0 microgram per milliliter (µg/mL) in the sera of subjects.
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 140 | 140 | 49 | 47
Participants | 139 | 137 | 48 | 45

20. Secondary Outcome: Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Antibody Concentrations
Description: Seroprotection status, defined as Anti-PRP antibody concentrations ≥ 0.15 µg/mL and ≥ 1.0 µg/mL
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 140 | 140 | 49 | 47
μg/mL | 26.001 [21.196 to 31.894] | 9.376 [7.941 to 11.071] | 25.758 [17.669 to 37.548] | 8.86 [6.87 to 11.427]

21. Secondary Outcome: Number of Subjects With Anti-diphtheria (Anti D) and Anti-tetanus Toxoids (Anti TT) Antibody Concentrations Equal to or Above 0.1 International Units Per Milliliter (IU/mL)
Description: Cut-off values assessed were greater than or equal to 0.1 International Units per milliliter (IU/mL) in the sera of subjects.
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 140 | 140 | 49 | 47
Participants
  Anti-diphtheria | 137 | 140 | 49 | 46
  Anti-tetanus: number analyzed (Participants) | 139 | 140 | 48 | 47
  Anti-tetanus | 139 | 140 | 48 | 47

22. Secondary Outcome: Anti-diphtheria (Anti-D) and Anti-tetanus Toxoids (Anti-TT) Antibody Concentrations
Description: Seroprotection status, defined as Anti-diphtheria toxoid or anti-tetanus toxoid antibody concentrations ≥ 0.1 IU/mL
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 140 | 140 | 49 | 47
IU/mL
  Anti-diphtheria | 1.735 [1.468 to 2.052] | 1.549 [1.356 to 1.771] | 1.252 [0.97 to 1.616] | 1.039 [0.786 to 1.375]
  Anti-tetanus: number analyzed (Participants) | 139 | 140 | 48 | 47
  Anti-tetanus | 5.195 [4.508 to 5.985] | 3.505 [3.148 to 3.904] | 3.476 [2.637 to 4.583] | 2.659 [2.091 to 3.381]

23. Secondary Outcome: Number of Subjects With Anti-Hepatitis B Surface Antigen (HBs) Antibody Concentrations Equal to or Above 10 Milli-International Units Per Milliliter (mIU/mL)
Description: Cut-off values assessed were greater than or equal to 10 milli-International Units per milliliter (mIU/mL) in the sera of subjects.
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 140 | 133 | 49 | 44
Participants | 127 | 132 | 44 | 44

24. Secondary Outcome: Anti-hepatitis B Surface Antigen (HBs) Antibody Concentrations
Description: Seroprotection status, defined as Anti-HBs antibody concentrations ≥ 10 mIU/mL
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 140 | 133 | 49 | 44
mIU/mL | 101.6 [79.7 to 129.5] | 756.7 [640.4 to 894.3] | 129.8 [83.3 to 202.1] | 792.2 [585.2 to 1072.2]

25. Secondary Outcome: Number of Subjects With Anti-polio Type 1, 2 and 3 Antibody Titers Equal to or Above (≥) 8
Description: Titers were expressed as geometric mean titres (GMTs).
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 124 | 120 | 44 | 41
Participants
  Anti-polio 1: number analyzed (Participants) | 123 | 120 | 44 | 40
  Anti-polio 1 | 120 | 120 | 40 | 40
  Anti-polio 2: number analyzed (Participants) | 124 | 116 | 43 | 41
  Anti-polio 2 | 124 | 115 | 43 | 41
  Anti-polio 3: number analyzed (Participants) | 120 | 108 | 38 | 39
  Anti-polio 3 | 116 | 107 | 32 | 39

26. Secondary Outcome: Anti-polio Type 1, 2 and 3 (Anti-Polio 1, 2 and 3) Antibody Titers
Description: Seroprotection status, defined as Anti-polio type 1, Anti-polio type 2 and Anti-polio type 3 antibody titers ≥ 8
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 124 | 120 | 44 | 41
Titers
  Anti-polio 1: number analyzed (Participants) | 123 | 120 | 44 | 40
  Anti-polio 1 | 641.5 [485.7 to 847.3] | 331.1 [269.5 to 406.8] | 373.7 [207.4 to 673.4] | 267.6 [187.5 to 381.8]
  Anti-polio 2: number analyzed (Participants) | 124 | 116 | 43 | 41
  Anti-polio 2 | 523.6 [436.9 to 627.5] | 276.8 [223 to 343.5] | 546.2 [370.5 to 805.2] | 303.5 [207.1 to 444.8]
  Anti-polio 3: number analyzed (Participants) | 120 | 108 | 38 | 39
  Anti-polio 3 | 204.5 [164.3 to 254.5] | 540.8 [433.7 to 674.3] | 101.9 [59.5 to 174.5] | 611.5 [449.4 to 832.2]

27. Secondary Outcome: Number of Subjects With Anti-Bordetella Pertussis (Anti-BPT) Antibody Concentrations Equal to or Above 15 ELISA Unit Per Milli-liter (EL.U/mL) (Seropositivity)
Description: Cut-off values assessed were greater than or equal to 15 ELISA unit per milli-liter (EL.U/mL) in the sera of subjects seronegative before vaccination.
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 138 | 133 | 48 | 45
Participants | 137 | 126 | 47 | 42

28. Secondary Outcome: Anti-Bordetella Pertussis (Anti-BPT) Antibody Concentrations
Description: Seropositivity status, defined as Anti-BPT antibody concentrations ≥ 15 EL.U/mL.
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 128 | 119 | 46 | 41
EL.U/mL | 72.465 [65.787 to 79.82] | 53.481 [47.215 to 60.579] | 77.175 [64.433 to 92.435] | 60.003 [46.394 to 77.604]

29. Secondary Outcome: Number of Subjects With Vaccine Response to Bordetella Pertussis
Description: Vaccine response to B. pertussis;defined as appearance of antibodies in subjects initially seronegative (S-) (i.e., concentrations < 15 EL.U/mL) or at least maintenance of pre-vaccination antibody concentrations in subjects who were initially seropositive (S+) (i.e., with concentrations ≥ 15 EL.U/mL).
Time Frame: One month after the administration of the 3rd vaccine dose of Tritanrix™-HepB/Hiberix™ + Polio Sabin™ or Poliorix™
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
Number analyzed (Participants) | 128 | 119 | 46 | 41
Participants
  S- | 127 | 112 | 46 | 38
  S+: number analyzed (Participants) | 9 | 14 | 2 | 4
  S+ | 9 | 12 | 1 | 2

ADVERSE EVENTS:
Time Frame: Solicited AEs: Within 4 day (Days 0-3) after each dose and across doses; Unsolicited AEs: Within 31 days (Days 0-30) after each vaccination. SAEs: From study Day 0 until the 6-month extended safety follow-up
Arm/Group | Synflorix 1 Group | Synflorix 2 Group | Prevenar 1 Group | Prevenar 2 Group
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/303 | 0/100 | 0/103
Serious Adverse Events (participants affected / at risk) | 16/300 | 52/303 | 4/100 | 19/103
Other Adverse Events (participants affected / at risk) | 296/300 | 300/303 | 95/100 | 98/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix 1 Group (N=300) | Synflorix 2 Group (N=303) | Prevenar 1 Group (N=100) | Prevenar 2 Group (N=103)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Double ureter (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 14 (16) | 0 (0) | 2 (2)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 9 (9) | 2 (2) | 2 (2)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7) | 8 (8) | 1 (1) | 3 (3)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix 1 Group (N=300) | Synflorix 2 Group (N=303) | Prevenar 1 Group (N=100) | Prevenar 2 Group (N=103)
Bronchitis (Infections and infestations) | 9 (9) | 6 (6) | 0 (0) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 140 (231) | 79 (152) | 39 (65) | 64 (99)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 7 (10) | 0 (0) | 8 (9)
Erythema (Skin and subcutaneous tissue disorders) | 221 (420) | 265 (360) | 67 (124) | 91 (195)
Gastroenteritis (Infections and infestations) | 17 (19) | 3 (3) | 7 (7) | 0 (0)
Haematoma (Vascular disorders) | 11 (11) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 258 (590) | 289 (732) | 82 (170) | 93 (221)
Nasopharyngitis (Infections and infestations) | 0 (0) | 10 (14) | 0 (0) | 4 (4)
Pain (General disorders) | 258 (599) | 86 (193) | 82 (175) | 89 (182)
Pharyngitis (Infections and infestations) | 4 (4) | 17 (18) | 2 (2) | 3 (4)
Pyrexia (General disorders) | 255 (543) | 262 (542) | 88 (187) | 77 (155)
Rhinitis (Infections and infestations) | 38 (42) | 39 (43) | 7 (10) | 9 (9)
Somnolence (Nervous system disorders) | 184 (346) | 256 (547) | 56 (95) | 85 (173)
Swelling (General disorders) | 174 (324) | 226 (467) | 42 (93) | 75 (160)
Upper respiratory tract infection (Infections and infestations) | 84 (97) | 16 (17) | 25 (31) | 12 (13)
Urinary tract infection (Infections and infestations) | 0 (0) | 8 (8) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 11 (11) | 1 (1) | 4 (4) | 0 (0)
Viral rhinitis (Infections and infestations) | 15 (16) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.